CLINICAL TRIAL: NCT02834975
Title: Phase II Single Arm Study of Combination Pembrolizumab, Paclitaxel, and Carboplatin in Patients With Advanced Stage Ovarian, Fallopian Tube, or Peritoneal Carcinoma Receiving Neoadjuvant Chemotherapy
Brief Title: Pembrolizumab, Paclitaxel, and Carboplatin in Patients With Advanced Stage Epithelial Ovarian Cancer (EOC).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: University of Miami (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Abdulrahman Sinno, MD, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160477
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Fallopian Tube Cancer; Peritoneum Cancer; Epithelial Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, Paclitaxel + Carboplatin (Experimental): The following therapy will be administered during each 21-day cycle for a maximum of eight (8) cycles:
  * Pembrolizumab 200mg intravenously (IV);
  * Paclitaxel 175 mg/m2 IV in a neoadjuvant setting (NACT);
  * Paclitaxel same as NACT, OR 80 mg/m2 IV dose dense option in an adjuvant setting (ACT);
  * Carboplatin IV area under the curve (AUC) of 6.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab on Day 1 of each cycle.
  Other Names: Keytruda; MK-3475
Drug: Paclitaxel — * NACT: Paclitaxel on Day 1 of each cycle;
  * ACT: Paclitaxel same as NACT OR; dose-dense option weekly per protocol.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin IV on Day 1 of each cycle.

SUMMARY:
The investigators hypothesize that tumor cell killing by cytotoxic chemotherapy exposes the immune system to high levels of tumor antigens.The combination of Paclitaxel/Carboplatin and Pembrolizumab may result in deeper and more durable responses compared with standard chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. No prior treatment for primary advanced (Stage III or IV) high grade epithelial ovarian, primary peritoneal, or fallopian tube carcinoma such as irradiation, chemotherapy, hormonal therapy, immunotherapy, investigational therapy, and/or other concurrent agents or therapies.
2. Patients must undergo diagnostic laparoscopy for disease assessment for tissue biopsies to confirm diagnosis with planned interval tumor reductive surgery after completion of 3-4 cycles of treatment. For those not medically fit to undergo laparoscopy, as determined by the Investigator. (interventional radiology) IR-guided core biopsies may be used.
3. Patients must be appropriate candidates for planned neoadjuvant chemotherapy (NACT) with combination carboplatin and paclitaxel given intravenously (IV) every 3 weeks ( IV Q3W).
4. Tissue from an archival sample or newly obtained core or excisional biopsy of a tumor lesion.
5. Age ≥ 18 years.
6. Life expectancy > 3 months.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
8. Patients must have normal organ and marrow function as defined below:

   * Hematologic

     * Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL).
     * Platelets ≥ 100,000 / mcL.
     * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or Erythropoietin (EPO) dependency
   * Renal

     * Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR
     * Measured or calculated a creatinine clearance ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl). Creatinine clearance should be calculated per institutional standard.
   * Hepatic

     * Serum total bilirubin ≤ 1.5 X ULN OR
     * Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
     * Aspartate transaminase (AST/SGOT) and Alanine transaminase (ALT/SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases.
     * Albumin > 2.5 mg/dL
   * Coagulation

     * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
     * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
9. Negative urine or serum pregnancy ≤ 72 hours (i.e. 3 days) prior to receiving the first dose of study medication if not surgically sterilized. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (have not been surgically sterilized or have not been without menses for > 1 year) should be willing to use 2 methods of birth control at the same time or be surgically sterile, or abstain from heterosexual activity for the course of the study and at least 120 days after the last study dose.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who are currently in or have participated in a study of an investigational agent or used an investigational device within 4 weeks of the first dose of treatment.
2. Histology showing mucinous or low grade epithelial ovarian cancer.
3. Patients who will not be likely to undergo IDS either secondary to performance status or sites of disease. If at the time of surgery, the patient is deemed to be surgically resectable to no gross residual, the patient will not be eligible for the study.
4. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to study treatment.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has received prior therapy with an anti-PD1, anti-PDL1, anti-CD137, anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) or anti-PDL2 agent.
7. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
9. Prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to previously administered event. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for this study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
11. Has active autoimmune disease that has required systemic treatment in the past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
13. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
14. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Received live vaccine within 30 days prior to the first dose of study treatment. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.
17. Patient has active bacillus tuberculosis (TB).
18. Patient with known hypersensitivity to pembrolizumab or any of its excipients (inactive ingredients).
19. Patient receiving concurrent additional biologic therapy.
20. Any other serious medical or psychiatric illness/condition likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huang, MD, MS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab, Paclitaxel + Carboplatin: The following therapy will be administered during each 21-day cycle for a maximum of eight (8) cycles:
  * Pembrolizumab 200mg intravenously (IV);
  * Paclitaxel 175 mg/m2 IV in a neoadjuvant setting (NACT);
  * Paclitaxel same as NACT, OR 80 mg/m2 IV dose dense option in an adjuvant setting (ACT);
  * Carboplatin IV area under the curve (AUC) of 6.
  Pembrolizumab: Pembrolizumab on Day 1 of each cycle.
  Paclitaxel: - NACT: Paclitaxel on Day 1 of each cycle;
  - ACT: Paclitaxel same as NACT OR; dose-dense option weekly per protocol.
  Carboplatin: Carboplatin IV on Day 1 of each cycle.
Period: Overall Study
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
Started | 26
Completed | 21
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Objective Response Rate (pORR) in Participants Receiving Protocol Therapy
Description: The pORR will be calculated as the percentage of participants with pathologic complete response (pCR) and pathologic partial response (pPR) overall as best response. For this protocol, pathologic complete response (pCR) will be defined as no residual macroscopic or (viable) microscopic disease. Pathologic partial response (pPR) will be defined as the presence of residual (viable) microscopic tumor, and the size of the largest focus will be provided for possible outcome correlation.
Time Frame: Up to 48 months
Population: Participants who received at least one dose of pembrolizumab in combination with paclitaxel and carboplatin will have tissue collected at baseline and at the time interval debulking surgery (IDS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
Number analyzed (Participants) | 25
percentage of participants | 60 [38.7 to 78.9]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is measured from date of start of treatment to the earliest occurrence of any of the following events: documented disease progression or death from any cause. Patients who are alive and progression-free will be censored at the date of last documented progression-free status which is the date of last tumor assessment according to RECIST v1.1.
Time Frame: Up to 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
Number analyzed (Participants) | 26
months | 22.5 [11.9 to NA] — Insufficient number of participants with disease progression.

3. Secondary Outcome: Number of Participants Experiencing Treatment-related Toxicity
Description: Safety and tolerability of the intervention will be reported as the number of participants experiencing treatment-related toxicity including serious adverse events (SAEs) and adverse events (AEs), as assessed by treating physician. Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0, per physician discretion.
Time Frame: Up to 48 Months
Population: All participants who received at least one dose of pembrolizumab in combination with paclitaxel and carboplatin.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
Number analyzed (Participants) | 26
Participants
  All Treatment-related SAEs | 3
  Grade 3 or higher treatment-related SAEs | 1
  All Treatment-related AEs (excluding SAEs) | 23
  Grade 3 or higher treatment-related AEs (excluding SAEs) | 10

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Pembrolizumab, Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 11/26
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab, Paclitaxel + Carboplatin (N=26)
Immune system disorder, other (Immune system disorders) | 1 (1) — Nephritis
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab, Paclitaxel + Carboplatin (N=26)
Anemia (Blood and lymphatic system disorders) | 9 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (13)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder, other (Gastrointestinal disorders) | 1 (1) — Flatus per vagina
Gastrointestinal disorder, other (Gastrointestinal disorders) | 1 (1) — H Pylory infection
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 14 (18)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 15 (21)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) — Bacteremia. Secondary to urinary tract infection (UTI)
Papulopustular rash (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 2 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 2 (5)
Cholesterol high (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (24)
Platelet count decreased (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Investigations) | 3 (3)
Hyperglycemia (Investigations) | 3 (3)
Hyponatremia (Investigations) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (4)
Neuralgia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (10)
Stroke (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Restlessness (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (15)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 1 (1) — Superficial Skin Separation
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (4)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02834975/Prot_SAP_000.pdf